CLINICAL TRIAL: NCT02655003
Title: TIME - Targeted Interdisciplinary Model for Evaluation and Treatment of Neuropscyhiatric Symptoms
Brief Title: Targeted Interdisciplinary Model for Evaluation and Treatment of Neuropscyhiatric Symptoms
Acronym: TIME
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Sykehuset Innlandet HF (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 150333
Record Dates: First submitted 2016-01-06; First posted 2016-01-13 (Estimated); Last update posted 2017-02-15 (Actual); Status verified 2016-10

CONDITIONS: Dementia
Keywords: behavioral symptoms; psychological symptoms; dementia; neuropsychiatric symptoms
MeSH Terms: conditions — Dementia; Behavioral Symptoms | interventions — Time

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- INH (Intervention Nursing Homes) (Experimental): TIME consists of a manual based multicomponent program which includes a rigorous assessment, the treatment, and the evaluation of NPS. The staff, physicians and nursing home managers in the intervention nursing homes will receive a one-day education program. Three nurses from each unit will receive further education including practical and theoretical training for three hours.
  Interventions: Other: TIME
- CNH (Control Nursing Homes) (Active Comparator): A brief two hours education-only intervention about dementia and NPS will be given to the staff in for the control nursing homes (CNH). The staff and physicians in the control nursing homes continue practice as usual.
  Interventions: Other: Education-only intervention

INTERVENTIONS:
Other: TIME
  Other Names: Targeted Interdisciplinary Model for Evaluation and treatment of neuropsychiatric symptoms
  Arms: INH (Intervention Nursing Homes)
Other: Education-only intervention — The staff and physicians in the control nursing homes will receive a 2 hours education session about dementia and neuropsychiatric symptoms
  Arms: CNH (Control Nursing Homes)

SUMMARY:
Almost all people who suffer from dementia experience neuropsychiatric symptoms (NPS) in the course of the disease. TIME (Targeted Interdisciplinary Model for Evaluation and treatment of neuropsychiatric symptoms) is a multicomponent intervention based on the theoretical framework of cognitive behavioral therapy (CBT). The TIME trial is designed to assess the effects of TIME on NPS in nursing homes patients with dementia and the implementation process at staff and organization level.

DETAILED DESCRIPTION:
TIME (Targeted Interdisciplinary Model for Evaluation and treatment of neuropsychiatric symptoms) is a multicomponent intervention based on the theoretical framework of cognitive behavioral therapy (CBT).The TIME trial includes a three months cluster randomized trial in 36 nursing homes with 164 participants with dementia and a high level of agitation. Each nursing home defines a cluster and will be randomized to receive either the intervention with TIME or a brief two hours education-only intervention about dementia and NPS for the control group. TIME consists of a manual based multicomponent program which includes a rigorous assessment, the treatment, and the evaluation of neuropsychiatrc symptoms (NPS). The staff, physicians and nursing home managers receive a one-day education. Three nurses from each unit will receive further education including practical and theoretical training for three hours. Measurements at patient level are taken at baseline prior to randomization and at eight and twelve weeks. The primary outcome measure is agitation. Mixed methods will be used to follow, measure and explore the implementation process and the effect at individual staff level and at organization level.

ELIGIBILITY:
Inclusion Criteria:

1. Clinical Dementia Rating scale (CDR) 1 or higher.
2. Moderate to high grade of agitation defined by the NPI-NH agitation item as equal to or above six points.
3. Planned long-term stay in the nursing home, and a minimum of two weeks stay in the nursing home before inclusion.

Exclusion Criteria:

1.Terminal phase (life expectancy less than 4-6 weeks)

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 229 (Actual)
Dates: Start 2016-01-07 (Actual); Primary Completion 2016-07-01 (Actual); Study Completion 2016-07 (Actual)

PRIMARY OUTCOMES:
NPI-NH agitation/aggression | 8 weeks and 12 weeks
  The primary outcome measure is change from baseline of agitation and aggression as defined by the Neuropsychiatric Inventory Nursing Home Version (NPI-NH) item agitation/aggression.

SECONDARY OUTCOMES:
NPI-NH all separate items | 8 weeks and 12 weeks
  The change from baseline of the remaining 11 items in the.Neuropsychiatric Inventory Nursing Home Version (NPI-NH).
NPI-NH sub syndrome agitation | 8 weeks and 12 weeks
  The change from baseline of the NPI-NH sub syndrome agitation is defined as the sum of the items agitation/aggression, irritability, and disinhibition in the NPI-NH.
NPI-NH sub syndrome affective symptoms | 8 weeks and 12 weeks
  The change from baseline of the NPI-NH sub syndrome affective symptoms is defined as the sum of the items depression and anxiety in the in the NPI-NH.
NPI-NH sub syndrome psychosis | 8 weeks and 12 weeks
  The change from baseline of the NPI-NH sub syndrome psychosis is defined as the sum of the items hallucinations and delusions items in the in the NPI-NH.
NPI-10 NH sum score | 8 weeks and 12 weeks
  The change from baseline of the NPI-10 NH sum score is the sum of the first ten items in the Neuropsychiatrc Inventory Nursing Homes version
The NPI-NH caregiver occupational disruptiveness score | 8 weeks and 12 weeks
  In the Neuropsychiatric Inventory Nursing Home Version (NPI-NH) the caregiver must rate how disruptive they find each behavior or symptom on a five point scale. The outcome is the change from baseline.
CMAI | 8 weeks and 12 weeks
  The change from baseline in the Cohen-Mansfield Agitation Inventory (CMAI) within its 29 different types of agitation and the frequency at which they occur.
Lawton and Brody ADL scale | 8 weeks and 12 weeks
  The change from baseline in the The Lawton and Brody ADL scale which describes 6 domains of activity of daily living with a score from 1 to 5 where 1 means no need for help and 5 means significant need for assistance.
The Cornell scale for depression in dementia CSDD | 8 weeks and 12 weeks
  The change from baseline in The Cornell scale for depression which measures the frequency of symptoms of depression.
Drug usage | 8 weeks and 12 weeks
  The change in drug dosage from baseline: that is the use of psychotropic and analgesic medication both as given regularly and on demand. This will be assessed using a questionnaire.
Quality of life measured by the scale QUALID | 8 weeks and 12 weeks
  The change from baseline in quality of life which will be assessed by the scale QUALID: Quality of life in late-stage dementia scale disease.
General medical health using the General Medical Health Rating scale | 8 weeks and 12 weeks
  The change from baseline in general medical health will be assessed by using the General Medical Health Rating scale (GMHR)

CONTACTS AND LOCATIONS:
Overall Officials: Sverre Bergh, PhD, Principal Investigator — +4745679393
Locations (1):
- Centre for Old Age Psychiatric Research, Sykehuset Innlandet Hospital Trust, Ottestad, Norway

REFERENCES:
- [Derived] Myhre J, Lichtwarck B. How and why does it work? A video-based qualitative analysis of case conferences to reduce BPSD through the lens of Habermas's theory of communicative action. BMC Psychiatry. 2024 Jul 22;24(1):520. doi: 10.1186/s12888-024-05959-x. PMID 39039488
- [Derived] Lichtwarck B, Myhre J, Selbaek G, Kirkevold O, Rokstad AMM, Benth JS, Bergh S. TIME to reduce agitation in persons with dementia in nursing homes. A process evaluation of a complex intervention. BMC Health Serv Res. 2019 May 31;19(1):349. doi: 10.1186/s12913-019-4168-0. PMID 31151437
- [Derived] Lichtwarck B, Selbaek G, Kirkevold O, Rokstad AM, Benth JS, Myhre J, Nybakken S, Bergh S. TIME - Targeted interdisciplinary model for evaluation and treatment of neuropsychiatric symptoms: protocol for an effectiveness-implementation cluster randomized hybrid trial. BMC Psychiatry. 2016 Jul 12;16:233. doi: 10.1186/s12888-016-0944-0. PMID 27406242